CLINICAL TRIAL: NCT00491777
Title: Correlation Study of NMT's IQ2, NcIQ and Its' Predicate Technology, IQ101.
Brief Title: Correlation Research Study: IQ2, NcIQ and IQ101
Acronym: NMT-CT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Noninvasive Medical Technologies, Inc. (Industry)
Collaborators: University of Florida (Other); Shand's Medical Center (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NMT-IQ2/NcIQ
Record Dates: First submitted 2007-06-22; First posted 2007-06-26 (Estimated); Last update posted 2007-06-26 (Estimated); Status verified 2007-06

CONDITIONS: Heart Failure; Dyspnea; Hypertension; Pacemaker; Trauma
Keywords: Noninvasive; Hemodynamic; Monitoring; Critical Care; Swan-Ganz
MeSH Terms: conditions — Heart Failure; Dyspnea; Hypertension; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Noninvasive Hemodynamic Patient Monitor

SUMMARY:
The new NcIQ thoracic impedance monitor is based on the predicate device, the IQ101. The new model uses the same 3-dimensional signal averaging as the original device, but also include second radio frequency signal to permit the device to work "wirelessly", i.e., without electrode lead attachments to the patient. This study seeks to 1) validate the use of the new device and confirm the correlation of the IQ101 and NcIQ. 2) Evaluate the ease of the new device.

The new IQ2 thoracic impedance monitor is based on the predicate device, the IQ101. The new model uses the same 3-dimensional signal averaging as the original device, but with smaller housing and updated operating software. This study seeks to 1) Validate the use of the new device and confirm the correlation of the IQ101 and IQ2. 2) Compare the ease of the devices.

DETAILED DESCRIPTION:
The IQ101 is the first generation of the non invasive cardiograph. This device uses impedance to a micro-electric field passing from the electrodes. The NcIQ uses Radio frequencies and the same 3 dimensional signal averaging algorithm used in the IQ101 to generate hemodynamic data. The radio waves enables the device to work without the contact lead arrays used in the IQ2 and can take measurements without even contacting the patient, hence can be applied through clothing and is simple to apply. This makes the potential use by first responders a possibility. The device measures the change in the radio wave reflection during the cardiac cycle to estimate ardiac function. Specifically, it measures cardiac output, the amount of blood pumped per minute, and other hemodynamic parameters previously only measurable with invasive catheters. The data us used to generate a LIFESCORE and can measure and report dangerous trends to the caretaker. The device has a companion device to download the data for the hospital providers to create a seamless transfer of care. The new device uses technology similar to the previous generation machine but has been miniaturized, given updated operating system, and newer computer technology that helped make the device smaller, and faster. The underlying patented algorithm was not changed. Therefore, it is expected to provide the same degree of accuracy and precision as the predicate device.

The IQ101 is the first generation of the non invasive cardiograph. This device uses impedance to a micro-electric field passing from the electrodes. The device can use the impedance and the change in the impedance during the cardiac cycle to estimate thoracic fluid volumes and cardiac function. Specifically, it measures cardiac output, the amount of blood pumped per minute, and other hemodynamic parameters previously only measurable with invasive catheters. There are many studies documenting the device's performance. The new device uses the same technology but has been modernized with updated operating system, and newer computer technology that helped make the device smaller, and faster. The device has also been redesigned to make operator use simpler and reduce the number wires involved. The underlying patented algorithm was not changed. Therefore, it is expected to provide the same degree of accuracy and precision as the predicate device with simplified user interface and lighter, smaller, more portable housing to improve ease of use.

ELIGIBILITY:
Inclusion criteria:

* Age - 18-80 years
* Weight - 80-300 pounds
* Height - 5.0 feet - 6feet 4 inches Exclusion Criteria
* Ongoing medical emergency or acute medical illness
* NcIQ or ECG electrode adhesive allergy or sensitivity

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-06; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
A direct correlation between output parameters of IQ2/NcIQ to IQ101

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Ferguson, MD, Study Chair — Shand's Hospital; Joseph A Tyndall, MD, Principal Investigator — Shand's Hospital; David Seaberg, MD, Study Director — Shand's Hospital